CLINICAL TRIAL: NCT07337824
Title: Comparison of Deep Neck Flexor Strengthening and Motor Learning-Based Neuroplasticity Training for Forward Head Posture
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Nimra Shahid
Record Dates: First submitted 2026-01-01; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Forward Head Posture
Keywords: Craniovertebral angle; Deep neck flexor strength; Proprioception; Neuroplasticity training; Motor learning

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental interventional group A (Deep neck flexor strengthening) (Experimental): * Chin tuck exercises
  * Isometric cervical flexion using gentle resistance
  * Prone head lift exercises
  Interventions: Other: Deep neck flexor strengthening
- Experimental :interventional group B ( Motor learning based neuroplasticity training) (Experimental): Task specific postural training using proprioceptive feedback, progressive balance and coordination and static and dynamic postural control tasks under different environmental conditions.
  Interventions: Other: Motor learning based neuroplasticity training

INTERVENTIONS:
Other: Deep neck flexor strengthening — Chin tuck exercises, Isometric cervical flexion using gentle resistance, Prone head lift exercises. Frequency: 3 sessions per week, Duration: 4 weeks (12 sessions total).
  Arms: Experimental interventional group A (Deep neck flexor strengthening)
Other: Motor learning based neuroplasticity training — Task-specific postural training using visual (laser), auditory (metronome), and proprioceptive feedback. Progressive balance and coordination exercises under varying environmental conditions. Static and dynamic postural control tasks with intertrial variability. Frequency: 3 sessions per week, Duration: 4 weeks (12 sessions total)
  Arms: Experimental :interventional group B ( Motor learning based neuroplasticity training)

SUMMARY:
The aim of this randomized clinical trial is to compare the effects of deep neck flexor strengthening and motor learning-based neuroplasticity training on craniovertebral angle, deep neck flexor strength, proprioception, and symptom recurrence in individuals with forward head posture (FHP).

The study will be conducted at Riphah International University, Gulberg Green Campus. A total of 74 participants with forward head posture will be recruited using non-probability convenience sampling and randomly allocated into two groups (37 participants per group). Group A will receive deep neck flexor strengthening exercises, while Group B will receive motor learning-based neuroplasticity training. Both groups will undergo three sessions per week for four weeks. Assessments will be performed at baseline, post-intervention, and at one-month follow-up to assess symptom recurrence. Data will be analyzed using SPSS version 27.

DETAILED DESCRIPTION:
Forward head posture is a prevalent postural abnormality characterized by anterior translation of the head relative to the cervical spine. It is commonly observed among university students and young adults due to prolonged smartphone use, computer work, and sedentary lifestyles. Persistent FHP leads to muscular imbalance, weakness of the deep neck flexors, altered proprioception, and impaired neuromuscular control, often resulting in neck pain and functional limitations.

Deep neck flexor strengthening targets the longus colli and longus capitis muscles to restore cervical alignment and improve segmental stability. These exercises aim to correct muscular imbalances by enhancing endurance and motor control of the cervical stabilizers.

Motor learning-based neuroplasticity training is an emerging rehabilitation approach that emphasizes sensorimotor integration, task-specific training, and multisensory feedback. This approach facilitates cortical reorganization and re-establishment of disrupted cortico-spinal and cortico-subcortical pathways through repetitive, goal-oriented motor tasks. By integrating visual, auditory, and proprioceptive feedback, neuroplasticity-based training enhances postural awareness, motor planning, and long-term postural correction.

Despite evidence supporting both interventions individually, limited research has directly compared their effectiveness across postural, neuromuscular, and proprioceptive outcomes, particularly with respect to symptom recurrence. This study seeks to address this gap.

Previous studies have demonstrated that deep neck flexor strengthening significantly improves craniovertebral angle, reduces neck pain, and enhances cervical stability in individuals with forward head posture. Cervical stabilization programs have also shown positive effects on proprioception and neck repositioning accuracy.

Recent randomized controlled trials investigating motor learning-based neuroplasticity approaches have reported improvements in postural control, proprioception, and functional movement patterns through experience-dependent cortical plasticity. However, systematic reviews highlight inconsistent evidence regarding the superiority of strengthening exercises over motor learning-based interventions, with limited comparative trials and short-term follow-up.

Furthermore, evidence related to symptom recurrence and long-term sustainability of postural correction remains scarce. Therefore, a direct comparison of these two interventions is warranted.

ELIGIBILITY:
Inclusion Criteria:

* University students aged 19-25 years
* Both genders
* Forward head posture with craniovertebral angle < 50°

Exclusion Criteria:

* History of cervical spine injury or surgery
* Chronic neck pain or recent therapy within six months.
* Diagnosed with neurological, musculoskeletal, or visual disorders affecting posture.

Ages: 19 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-01-20 (Estimated)

PRIMARY OUTCOMES:
Craniovertebral Angle (CVA) | Baseline to 4 weeks
  Measured using digital photogrammetry and analyzed with software (e.g., Kinovea) to quantify forward head posture severity.

SECONDARY OUTCOMES:
Deep Neck Flexor Strength | Baseline to 4 weeks
  Assessed using the Deep Neck Flexor Endurance Test. It is performed in the supine line position with the chin hold and head off the couch and ask the patient to hold the position. The time of the hold will be recorded.
Cervical Proprioception | Baseline to 4 weeks
  Measured using the Cervical Joint Repositioning Error Test with laser-guided repositioning.
Deep Neck Extensor Strength | Baseline to 4 weeks
  Assessed using the Deep Neck Extensor Endurance Test. It is performed in the prone line position with the chin hold and head off the couch and ask the patient to hold the position. The time of the hold will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Aisha Razzaq, PHD*, Principal Investigator — Riphah International University
Locations (1):
- Riphah Postgraduate Lab, Riphah INternational University, Islamabad, Capital, Pakistan

IPD SHARING:
Plan to Share IPD: No